CLINICAL TRIAL: NCT05201716
Title: Turkish Validity and Reliability of the UW Concerns About Pain Scale
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Saracoglu, Asst. Prof., Kutahya Health Sciences University
Other Study IDs: KutahyaHSU2
Record Dates: First submitted 2022-01-09; First posted 2022-01-21 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Chronic Low-back Pain
Keywords: Concerns

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brief Summary:

The aim of this study was to determine the Turkish validity and reliability of ''UW Concerns About Pain Scale'' developed by Dr. Amtmann.

DETAILED DESCRIPTION:
Chronic pain is a common condition, affecting an estimated 20% of people worldwide. The biopsychosocial model of chronic pain is the most current accepted approach to understanding the complexity of pain and disability. One of the most important psychosocial factors in this approach is pain-related self-efficacy, which is defined as the individual's confidence in their ability to tolerate pain and participate in daily activities despite pain. The aim of this study is to determine the Turkish version, validity, and reliability of ''UW Concerns About Pain Scale''. 60 people with chronic low back pain will include in the study. In order to determine the reliability of the scale, the intraclass correlation coefficient (ICC) will be used to determine the level of the relationship between the results of the first and second measurements. Cronbach's alpha coefficient will be used for the homogeneity of the questions in the scale. For construct validity, the correlation coefficient will be used to determine the agreement between the Turkish version of Pain catastrophizing scale and, Turkish version of "Fear Avoidance Beliefs Questionnaire" and The ''UW Concerns About Pain Scale''.

ELIGIBILITY:
Inclusion Criteria:

1. To be between 18-65 years old
2. Having a complaint of low back pain for at least 6 months
3. Low back pain severity to be 3 points or above according to the Numerical Graded Pain Scale.

Exclusion Criteria:

1. Using antidepressant-derived drugs
2. Having a history of spinal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with Chronic low back pain
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
UW Concerns About Pain | 8 minutes
  The UW Concerns About Pain is intended measure an individual's level of pain catastrophizing. We will use to 8 item form, in study.

SECONDARY OUTCOMES:
Turkish version of Pain Catastrophizing Scale (PCS) | 10 minutes
  PCS was developed by Sullivan et al. in order to identify the catastrophic thoughts or feelings of the patients about the pain and ineffective coping strategies.The scale is a Likert-type self-assessment scale consisting of 13 items.Each item is scored between 0-4 points.The total score ranges from 0 to 52.High scores indicate a high level of catastrophizing.
Turkish version of "Fear Avoidance Beliefs Questionnaire" | 10 minutes
  FABQ was developed Waddell et al. in 1993. FABQ consists of 16 questions and 2 parts. While the first part of the scale evaluates attitudes about physical activities, the second part evaluates attitudes about occupational work. Scoring of the questionnaire is done with a 7-point Likert type scale. The Physical Activity section is scored between 0-24 and the labor section is scored between 0-36. A high score in KKTS indicates an increased level of fear-avoidance attitudes related to low back pain.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail SARACOGLU, PhD, Study Director — Kutahya Health Sciences University; Cihan Caner AKSOY, PhD, Principal Investigator — Kutahya Health Sciences University; Lütfiye AKKURT, MSc, Principal Investigator — Kutahya Health Sciences University; Hasan Hüseyin GÖKPINAR, MD, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)